CLINICAL TRIAL: NCT00004828
Title: Liothyronine in Children With Single Ventricle Congenital Cardiac Malformations Undergoing the Fontan Procedure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Children's Hospital and Health Center (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13357; CHSD-585; CHSD-FDR001195
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-06

CONDITIONS: Tricuspid Atresia; Heart Defects, Congenital
Keywords: cardiovascular and respiratory diseases; heart defects; rare disease
MeSH Terms: conditions — Tricuspid Atresia; Heart Defects, Congenital; Respiratory Tract Diseases; Rare Diseases

INTERVENTIONS:
Drug: liothyronine I 131

SUMMARY:
OBJECTIVES: I. Determine the pharmacokinetics of exogenous liothyronine administered in children undergoing the modified Fontan procedure.

II. Determine the liothyronine supplementation dose that counters the fall in serum liothyronine concentrations and provides the greatest potential myocardial benefit after the modified Fontan procedure.

III. Evaluate the potential toxicity of exogenous liothyronine administered in children undergoing a modified Fontan procedure.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, placebo controlled, dose escalation study.

Initially, patients are randomized to receive either 1 of 3 different dosages of liothyronine or placebo after undergoing the Fontan procedure. If no unacceptable toxicity is observed in this group, a third dose level of liothyronine is added to the randomization. A total of 7 patients are enrolled at each dose level. All randomized study drugs are administered by continuous infusion over 1 hour after surgery.

Cardiac function is assessed 5 days after surgery.

ELIGIBILITY:
* Single ventricle congenital cardiac malformation
* Must undergo modified Fontan procedure
* No concurrent medications known to interfere with thyroid metabolism including propranolol and amiodarone
* No hepatic dysfunction
* No renal dysfunction
* No pre-existing thyroid dysfunction

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28
Dates: Start 1994-12; Study Completion 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mainwaring, Study Chair — Children's Hospital and Health Center